CLINICAL TRIAL: NCT01197339
Title: Hybrid Model of Vocal Inflammation and Tissue Mobilization
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH); McGill University (Other); Purdue University (Other)
Responsible Party: Principal Investigator, Kittie Verdolini Abbott, Professor, University of Pittsburgh
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Basic Science
Other Study IDs: DC008290; 5R01DC008290 (NIH)
Record Dates: First submitted 2010-09-07; First posted 2010-09-09 (Estimated); Last update posted 2016-01-25 (Estimated); Status verified 2016-01

CONDITIONS: Acute Phonotrauma
Keywords: acute phonotrauma; computer modeling; resonant voice; breathy voice; voice rest; relaxation
MeSH Terms: interventions — Meditation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- treatment (Experimental)
  Interventions: Behavioral: resonant voice; Behavioral: Breathy voice; Behavioral: Relaxation exercise; Behavioral: Resonant voice and relaxation exercise
- Controls (Sham Comparator)
  Interventions: Behavioral: voice rest

INTERVENTIONS:
Behavioral: resonant voice — A 4-hr resonant voice exercise will be prescribed to subjects following vocal loading.
  Arms: treatment
Behavioral: voice rest — A 4-hr voice rest will be prescribed to subjects following vocal loading.
  Arms: Controls
Behavioral: Breathy voice — A 4-hr breathy voice exercise will be prescribed to subjects following vocal loading.
  Arms: treatment
Behavioral: Relaxation exercise — A 4-hr relaxation exercise will be prescribed to subjects following vocal loading.
  Other Names: meditation
  Arms: treatment
Behavioral: Resonant voice and relaxation exercise — A 4-hr resonant voice and relaxation exercise will be prescribed to subjects following vocal loading.
  Other Names: Resonant voice and meditation exercise
  Arms: treatment

SUMMARY:
The purpose of this study is to generate a technology that will allow clinicians to prescribe behavioral treatment that should optimize tissue healing for both acute and chronic phonotrauma. In this study, we propose to (1): establish a non-invasive methodology for estimating overall mechanical dose during phonation, and component metrics of phonatory mechanical dose (e.g., distance dose, energy dissipation dose and time dose) from high speed imaging data and aeromechanical modeling, for a range of vocal fold configurations (Experiment 1); (2): identify mathematical relations between treatment dose parameters, inflammatory state of the tissue and time-varying biological consequences in the tissue, up to 2 wk following acute phonotrauma (Experiment 2); (3): develop a hybrid physical-biological model of vocal fold inflammation and treatment to identify treatment modalities that should optimize post-traumatic wound healing at 2 wk, for a range of acute phonotraumatic conditions (Experiment 3-no human subject involved), and (4): provide a preliminary test of the hybrid treatment models' ability to predict idealized treatment outcome in human subjects, and calibrate the model as needed iteratively to achieve a match between predicted and obtained outcomes (Experiment 4).

ELIGIBILITY:
Inclusion Criteria:

* healthy females
* ages 18-40
* generally healthy
* normal hearing bilaterally at 20 dB to 8,000 Hz
* have ability to produce "resonant voice" during training as determined by the examiner perceptually
* Tolerate rigid and nasal endoscopy without anesthesia to the larynx nasal patency allowing for the passage of an endoscope unilaterally

Exclusion Criteria:

* Smoking within the past five yr
* Failing a hearing screening test
* Having current chronic voice problems
* Having current medications that are determined to possibly influence voice
* Having heightened gag reflex
* Having known or suspected allergy to anesthetics
* Pregnancy reported

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2010-09; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Biomarker levels in laryngeal secretion | up to 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Verdolini Abbott, Ph.D., Principal Investigator — University of Pittsburgh
Locations (1):
- Univesity of Pittsburgh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Result] Li NY, Abbott KV, Rosen C, An G, Hebda PA, Vodovotz Y. Translational systems biology and voice pathophysiology. Laryngoscope. 2010 Mar;120(3):511-5. doi: 10.1002/lary.20755. PMID 20025041